CLINICAL TRIAL: NCT06257043
Title: RECORD TAVR REGISTRY: Prospective, Multi-Center Registry of "Real World" Chinese Patients Undergoing Transcatheter Aortic Valve Replacement
Brief Title: Safety and Efficacy of Post-marketing Transcatheter Aortic Valves in "Real World" Chinese Patients
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Other Study IDs: RECORD TAVR REGISTRY
Record Dates: First submitted 2023-12-21; First posted 2024-02-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Disease Mixed
Keywords: Aortic Valve Disease; Real world; TAVR
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transcatheter aortic valve replacement — A total of 3000 consecutive patients with aortic valve disease undergoing TAVR will be enrolled at 30-50 centers. The devices used will be all post-market transcatheter aortic valves approved for use in China. Clinical follow-up will be conducted in the periprocedural and after aortic valve implantation at 1 month, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years
  Other Names: Transcatheter aortic valve implantation

SUMMARY:
The purpose of this prospective multi-center, observational registry in China is to collect clinical baseline, procedural, and follow-up data of all patients treated with TAVR in China and to evaluate short-, mid-, and long-term clinical outcome data of all post-marketing transcatheter valves. Each center will collect baseline and procedural data as well as clinical outcomes for up to 10 years.

DETAILED DESCRIPTION:
Aortic stenosis is the most clinically important valvular heart disease in the elderly, with severe aortic stenosis accounting for about 3.4%-5% of elderly patients. Patients with chest pain, congestive heart failure, or syncope who do not undergo surgical intervention have a poor prognosis, with a 1-year mortality rate as high as 50%. However, the high surgical risk of surgical valve replacement for elderly patients with multiple underlying diseases limits the use of surgical valve replacement, and the prognosis of high-risk surgical patients is poor. The PARTNER series of studies and the US CoreValve high-risk studies confirm that perioperative and postoperative adverse events in patients undergoing TAVR in surgical high-risk patients are comparable to those in surgical valve replacement. With technological advances, the indications for TAVR have been expanded from surgical high-risk to low to moderate-risk populations. Based on the PARTNER 3 and Evolut Low Risk studies, FDA approved the use of TAVR to treat low surgical risk patients with symptomatic severe aortic stenosis. Recently, TAVR has also been expanded to patients with aortic valve regurgitation.

With a population of 1.4 billion, China has a large number of patients with aortic valve disease, but the TAVR program was launched in 2010. No large-scale TAVR studies are available to validate the efficacy and safety of TAVR in the Chinese population. The morphological characteristics of valves in our patients bring great challenges to the operation and application of TAVR. However, through the efforts of Chinese experts and scholars, TAVR technology in China has developed rapidly, and various domestic valves with independent intellectual property have been marketed, bringing new opportunities for the promotion and application of TAVR in China. Domestic valves have been designed for the Chinese aortic valve anatomy, which is theoretically more suitable for the Chinese population. However, the efficacy and safety of these valves still need to be further confirmed in large clinical studies.

This multi-center registry study aims to evaluate the safety and efficacy of all post-marketing transcatheter valves in Chinese patients with aortic valve disease mixed. Investigators will collect baseline and procedural data, and evaluate the short-, mid-, and long-term clinical outcomes of TAVR in a large real-world population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with aortic valve disease are evaluated by the cardiac team and indicate TAVR therapy
2. Patients who understand the purpose of this study, voluntarily participate in the trial and sign the informed consent form

Exclusion Criteria:

1. Patients with aortic valve disease who have been evaluated by a cardiac team as unsuitable for TAVR
2. Patients who cannot tolerate the materials or medications associated with this study
3. Women who are pregnant or breastfeeding
4. Patients who participated in a clinical trial of another drug or medical device before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with aortic valve disease who are evaluated by the cardiac team for TAVR treatment
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2033-11-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Combined early safety and clinical efficacy outcomes as defined by the Valve Academic Research Consortium-3 (VARC-3) | 1 year
  Composed by all-cause mortality, all strokes, any hospitalization, myocardial infarction

SECONDARY OUTCOMES:
Combined early safety and clinical efficacy outcomes as defined by the Valve Academic Research Consortium-3 (VARC-3) | 30 days
  Composed by all-cause mortality, all strokes, any hospitalization, myocardial infarction, acute kidney injury, life-threatening or fatal bleeding, mild or greater prosthetic valve regurgitation, new permanent pacemaker implantation, conduction block and arrhythmia, vascular and access-related complications, structural cardiac complications, any other adverse events
Rate of technical success | at exit from procedure room
  Technical success
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the devicea or to a major vascular or access-related, or cardiac structural complication
Rate of device success | discharge or 30 days
  Device success
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient <20mmHg, peak velocity <3 m/s, Doppler velocity index >_0.25, and less than moderate aortic regurgitation)
Combined safety and clinical efficacy outcomes as defined by the Valve Academic Research Consortium-3 (VARC-3) | 2 years, 3 years, 4 years
  Composed by all-cause mortality, all strokes, any hospitalization, myocardial infarction, life-threatening or fatal bleeding, mild or greater prosthetic valve regurgitation, new permanent pacemaker implantation, conduction block and arrhythmia, any other adverse events
Combined safety and clinical efficacy outcomes as defined by the Valve Academic Research Consortium-3 (VARC-3) | 5 years and 10 years
  Composed by all-cause mortality, all strokes, any hospitalization, myocardial infarction, life-threatening or fatal bleeding, mild or greater prosthetic valve regurgitation, new permanent pacemaker implantation, conduction block and arrhythmia, structural valve deterioration, any other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D, Ph.D, Study Chair — Xijing Hospital; Rutao Wang, M.D, Ph.D, Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No